CLINICAL TRIAL: NCT02057679
Title: Extended Antibiotic Therapy in Postoperative of Laparoscopic Cholecystectomy Due to Acute Cholecystitis. Is it Necessary?
Brief Title: Extended Antibiotic Therapy in Postoperative of Laparoscopic Cholecystectomy in Acute Cholecystitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, MARTIN DE SANTIBAÑES, MD, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2111
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Acute Cholecystitis
Keywords: Acute cholecystitis.; Amoxicillin clavulanic
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Amoxicillin-Potassium Clavulanate Combination; Lactose

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Amoxicillin Clavulanic) (Active Comparator): Intake of active drug (Amoxicillin Clavulanic). 3 g per day divided into 3 oral intakes of 1 g each (2 pill of Amoxicillin Clavulanic every 8 hrs). This treatment will begin on postoperative day 1 for 5 days.
  Interventions: Drug: Amoxicillin clavulanic
- Placebo (Placebo Comparator): Intake of placebo (Lactose). 1 pill of the same characteristics as Amoxicillin clavulanic every 8 hs. This will begin on postoperative day 1 for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin clavulanic — 3 g per day divided into 3 oral intakes of 1 g each (2 pill of Amoxicillin Clavulanic every 8 hrs). This treatment will begin on postoperative day 1 for 5 days.
  Other Names: Optamox
  Arms: Group A (Amoxicillin Clavulanic)
Drug: Placebo — 1 pill of the same characteristics as Amoxicillin clavulanic every 8 hs. This will begin on postoperative day 1 for 5 days.
  Other Names: Lactose
  Arms: Placebo

SUMMARY:
Acute cholecystitis (AC) is a very common complication of cholelithiasis, encountered in 20% of symptomatic patients.

Nowadays laparoscopic cholecystectomy (LC) is the standard treatment in mild and moderates forms of diseases and antibiotic therapy in the postoperatory of these patients remains under discussion. However in the beginning, AC presents itself as an steril process, the obstruction of the cystic duct initiates a cascade of inflammation, ischaemia and necrosis, as well as bacterial proliferation within the gallbladder lumen. Bactibilia was a significant factor associated with total, as well as infectious, operative complications. Regarding this, for some authors, monotherapy with amoxicillin clavulanic (AMC) would be the best treatment after LC in patients with mild and moderate cholecystitis without intraoperative complications such as bile peritonitis, cholangitis, gallbladder perforation or abscess. In the other hand, others do not prescribe antimicrobial treatment after surgery in these selected patients.

There is controversy regarding the postoperative treatment with antibiotics in patients with mild and moderate cholecystitis and all the evidence about this topic.

Therefore, investigators decided to conduct a prospective randomized study in patients undergoing laparoscopic cholecystectomy for acute mild and moderate cholecystitis cancer. The patients will be randomized to receive AMC or placebo after surgery. With this study investigators intend to prove that are no clinical differences in postoperative outcomes between patients treated with AMC and placebo.

The primary aim of the trial is to assess that there are no benefits in the use of postoperative antibiotics in patients whit mild or moderate acute cholecystitis in whom a laparoscopic cholecystectomy was performed.

DETAILED DESCRIPTION:
Double blind randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years old
* Patients with diagnose of mild or moderate acute cholecystitis.
* Underwent laparoscopic cholecystectomy on Italian Hospital of Buenos Aires

Exclusion Criteria:

* They refuse to participate from the trial or the process of informed consent.
* Have known allergies or hypersensitivity to Mosapride or lactose (used for placebo).
* Patients with severe cholecystitis
* Patients with moderate cholecystitis who presents liver abscess, gallbladder abscess, cholangitis or bile peritonitis.
* Intraoperative findings like liver cancer, liver metastases, common bile duct stones or gallbladder carcinoma.
* Patients with conversion to laparotomy
* Previous treatment with antibiotics for more than five days.
* Patients with active oncological diseases, AIDS, diabetes, transplanted.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-02; Primary Completion 2017-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Incidence of infectious postoperative complications | 30 days
  Incidence of infectious postoperative complications in patients who underwent a laparoscopic cholecystectomy due to acute mild and moderate cholecystitis, with antibiotics or placebo

SECONDARY OUTCOMES:
Number of days of hospital stay or readmissions. | 30 days
  To evaluate hospital stay.
Number of surgical reinterventions or reoperations. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin de Santibañes, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Diego Giunta, MD, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Buenos Aires, Argentina

REFERENCES:
- [Background] Strasberg SM. Clinical practice. Acute calculous cholecystitis. N Engl J Med. 2008 Jun 26;358(26):2804-11. doi: 10.1056/NEJMcp0800929. No abstract available. PMID 18579815
- [Background] Yoshida M, Takada T, Kawarada Y, Tanaka A, Nimura Y, Gomi H, Hirota M, Miura F, Wada K, Mayumi T, Solomkin JS, Strasberg S, Pitt HA, Belghiti J, de Santibanes E, Fan ST, Chen MF, Belli G, Hilvano SC, Kim SW, Ker CG. Antimicrobial therapy for acute cholecystitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):83-90. doi: 10.1007/s00534-006-1160-y. Epub 2007 Jan 30. PMID 17252301
- [Background] Yildiz B, Abbasoglu O, Tirnaksiz B, Hamaloglu E, Ozdemir A, Sayek I. Determinants of postoperative infection after laparoscopic cholecystectomy. Hepatogastroenterology. 2009 May-Jun;56(91-92):589-92. PMID 19621660
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Yokoe M, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Gomi H, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Kiriyama S, Kimura Y, Tsuyuguchi T, Itoi T, Yoshida M, Miura F, Yamashita Y, Okamoto K, Gabata T, Hata J, Higuchi R, Windsor JA, Bornman PC, Fan ST, Singh H, de Santibanes E, Kusachi S, Murata A, Chen XP, Jagannath P, Lee S, Padbury R, Chen MF; Tokyo Guidelines Revision Committee. New diagnostic criteria and severity assessment of acute cholecystitis in revised Tokyo Guidelines. J Hepatobiliary Pancreat Sci. 2012 Sep;19(5):578-85. doi: 10.1007/s00534-012-0548-0. PMID 22872303
- [Background] Kanafani ZA, Khalife N, Kanj SS, Araj GF, Khalifeh M, Sharara AI. Antibiotic use in acute cholecystitis: practice patterns in the absence of evidence-based guidelines. J Infect. 2005 Aug;51(2):128-34. doi: 10.1016/j.jinf.2004.11.007. Epub 2005 Jan 20. PMID 16038763
- [Background] Grande M, Torquati A, Farinon AM. Wound infection after cholecystectomy. Correlation between bacteria in bile and wound infection after operation on the gallbladder for acute and chronic gallstone disease. Eur J Surg. 1992 Feb;158(2):109-12. PMID 1350211
- [Background] Galili O, Eldar S Jr, Matter I, Madi H, Brodsky A, Galis I, Eldar S Sr. The effect of bactibilia on the course and outcome of laparoscopic cholecystectomy. Eur J Clin Microbiol Infect Dis. 2008 Sep;27(9):797-803. doi: 10.1007/s10096-008-0504-8. Epub 2008 Mar 28. PMID 18369670
- [Derived] Pellegrini P, Campana JP, Dietrich A, Goransky J, Glinka J, Giunta D, Barcan L, Alvarez F, Mazza O, Sanchez Claria R, Palavecino M, Arbues G, Ardiles V, de Santibanes E, Pekolj J, de Santibanes M. Protocol for extended antibiotic therapy after laparoscopic cholecystectomy for acute calculous cholecystitis (Cholecystectomy Antibiotic Randomised Trial, CHART). BMJ Open. 2015 Nov 18;5(11):e009502. doi: 10.1136/bmjopen-2015-009502. PMID 26582405